CLINICAL TRIAL: NCT07114874
Title: A Global, Phase 3, Multicenter, Open-Label Study to Assess the Long-Term Safety and Tolerability of NBI-1117568 in Adults With Schizophrenia
Brief Title: NBI-1117568-SCZ3032: Long-Term Evaluation of NBI-1117568 in Adults With Schizophrenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-1117568-SCZ3032; 2025-521216-19-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-29; First posted 2025-08-11 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NBI-1117568 (Experimental): Participants will receive NBI-1117568 once daily (QD) orally for up to 36 months.
  Interventions: Drug: NBI-1117568

INTERVENTIONS:
Drug: NBI-1117568 — NBI-1117568 will be administered per schedule specified in the arm description.

SUMMARY:
This study will evaluate the long-term safety of NBI-1117568 in adults with schizophrenia.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a primary diagnosis of schizophrenia
* Participants taking prohibited medications, including antipsychotics, must discontinue before study participation
* Participant must reside in a stable housing situation

Key Exclusion Criteria:

* Participant has known hypersensitivity to any component of the formulation of NBI-1117568
* Participant has an unstable or poorly controlled medical condition or chronic disease
* Participant is considered by the investigator to be at imminent risk of suicide or injury to self or others
* Participant has a diagnosis of moderate or severe substance use disorder (with the exception of nicotine or caffeine dependence) within 6 months prior to screening
* Participant has a positive alcohol test or drug screen for disallowed substances
* Participant has a history of poor or suspected poor compliance in clinical research studies and/or in the investigator's opinion, the participant is not capable of adhering to the protocol requirements.

Note: Other protocol-specified inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (23):
- United States (23):
  - Neurocrine Clinical Site, Little Rock, Arkansas
  - Neurocrine Clinical Site, Culver City, California
  - Neurocrine Clinical Site, Garden Grove, California
  - Neurocrine Clinical Site, Pico Rivera, California
  - Neurocrine Clinical Site, Riverside, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, Sherman, California
  - Neurocrine Clinical Site, Torrance, California
  - Neurocrine Clinical Site, Hollywood, Florida
  - Neurocrine Clinical Site, Miami Lakes, Florida
  - Neurocrine Clinical Site, Atlanta, Georgia
  - Neurocrine Clinical Site, Decatur, Georgia
  - Neurocrine Clinical Sites, Peachtree Corners, Georgia
  - Neurocrine Clinical Site, Chicago, Illinois
  - Neurocrine Clinical Site, Gaithersburg, Maryland
  - Neurocrine Clinical Site, Watertown, Massachusetts
  - Neurocrine Clinical Site, St Louis, Missouri
  - Neurocrine Clinical Site, Marlton, New Jersey
  - Neurocrine Clincial Site, Staten Island, New York
  - Neurocrine Clinical Sites, The Bronx, New York
  - Neurocrine Clinical Sites, North Canton, Ohio
  - Neurocrine Clinical Site, Austin, Texas
  - Neurocrine Clinical Sites, Orem, Utah